CLINICAL TRIAL: NCT03306147
Title: Negating Opioid and Pain Actively Through Intervention
Acronym: NOPAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: Cardinal Health (Industry)
Responsible Party: Principal Investigator, Huy Le, Medication Safety/Pharmacy Quality Management Coordinator, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5170244
Record Dates: First submitted 2017-10-04; First posted 2017-10-10 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Pain; Chronic Pain; Opioid Use
Keywords: Pain; Opioid; Drug monitoring; Pain education
MeSH Terms: conditions — Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic pain or long-acting opioid use (Experimental): Education of pain and promotion of adjunct and non-pharmacologic alternative therapies will be completed to engage patients in assessing their pain and seeing the effectiveness of their treatment. Patients will receive 3 follow-up interventions: 2 phone calls with a pharmacist or student pharmacist at weeks 2 and 6, and a follow-up visit with a pain or primary care physician.
  Interventions: Behavioral: Pain education with follow up encounters

INTERVENTIONS:
Behavioral: Pain education with follow up encounters — Patient pain review, counseling and education by pharmacists and physicians in follow up encounters

SUMMARY:
Chronic pain is one of the most prevalent and debilitating medical conditions and opioid analgesics are a commonly prescribed class of medications in the United States. Opioid efficacy has been proven in terms of managing acute and chronic pain; however, opioid overdose deaths, addictions, and diversions have all continued to increase over the years. The purpose of this study is to increase patient engagement in pain management and education, and to decrease opioid use by 10% over the study period. This study will also help present opportunities for future studies to obtain insight regarding the chronic use of opioids.

DETAILED DESCRIPTION:
The institutional review board has approved this prospective single-center study at a large 900-bed academic university medical center. The electronic medical record system will identify 300 patients, who are at least 18 years of age, with a history of opioid use for 3 or more months, or who are currently prescribed and are using long-acting or extended release opioids. Procedures by student pharmacists, pharmacy residents, and pharmacists will include reviewing medical records and prescription drug monitoring programs for the use of opioids, evaluating baseline pain, quality of life, and satisfaction via questionnaires and assessment questions, and performing thorough medication consultations on current opioid regimens. Education of pain and promotion of adjunct and non-pharmacologic alternative therapies will be completed to engage patients in assessing their pain and seeing the effectiveness of their treatment. Patients will receive 3 follow-up interventions: 2 phone calls with a pharmacist or student pharmacist at weeks 2 and 6, and a follow-up visit with a pain or primary care physician. Opioid usage, pain, quality of life, and patient satisfaction will be assessed. The primary outcome measured will be a decrease in opioid usage in morphine milligram equivalents. Secondary outcomes include change in quality of life and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* history of opioid use for 3 or more months or
* currently prescribed and are using long-acting or extended release opioids

Exclusion Criteria:

* substance use
* oncology patients
* hematology patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Decrease in opioid prescription strength | Change in prescription strength between date of subject enrollment and 90 days after subject enrollment date
  Opioid usage will be measured by changes in prescription strength of morphine milligram equivalents

SECONDARY OUTCOMES:
Reduction in pain as evidenced by decrease in opioid daily dose | Change in daily opioid use between date of subject enrollment and 90 days after subject enrollment date
  Subject will keep a daily opioid calendar to track their opioid daily dose
Improvement in quality of life score as measured by the PEG pain screening tool by units on a scale | Change in quality of life score as measured by the PEG pain screening tool by units on a scale between date of subject enrollment and 90 days after subject enrollment date
  Survey will be administered by investigators and completed by the patients before and after the interventions

CONTACTS AND LOCATIONS:
Overall Officials: Huy Le, PharmD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No